CLINICAL TRIAL: NCT00892112
Title: Immunoglobulin Therapy for Patients With Idiopathic Cardiomyopathy and Endomyocardial Parvovirus B19 Persistence - a Prospective, Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Intravenous Immunoglobulin (IVIg) for Parvovirus B19(PVB19) Mediated Cardiomyopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD2009.01
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Diseases; Parvovirus B19, Human
Keywords: Immunoglobulins, Intravenous; Cardiomyopathies; Parvo B19, Human
MeSH Terms: conditions — Cardiomyopathies | interventions — Immunoglobulins, Intravenous; Plasma Substitutes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous immunoglobulins (Active Comparator): IV, 40 ml/kg over 4 days
  Interventions: Drug: Intravenous Immunoglobulins
- plasma volume expander Albuman (Placebo Comparator): IV, 40 ml/kg over 4 days
  Interventions: Drug: plasma volume expander

INTERVENTIONS:
Drug: Intravenous Immunoglobulins — 2 gr/kg body weight of intravenous immunoglobulin product Nanogam® administered as 0.5 gr/kg IV over a period of 6 hours on each of 4 consecutive days
  Other Names: Nanogam
  Arms: intravenous immunoglobulins
Drug: plasma volume expander — 10 ml/kg BW will be administrated on four consecutive days.
  Other Names: G.P.O. ("Gepasteuriseerde Plasma-eiwit Oplossing"); Albuman 40 g/l
  Arms: plasma volume expander Albuman

SUMMARY:
A prospective randomized double-blind placebo-controlled trail to investigate the effect of high doses of IVIg on cardiac functional capacity and virus presence in a subgroup of patients with chronic symptomatic ICM and a high PVB19 load in the heart.

DETAILED DESCRIPTION:
Rationale: Parvovirus B19 (PVB19) persistence in the heart has been associated with progressive cardiac dysfunction and evolution to idiopathic cardiomyopathy.

Objective: A controlled trial to investigate whether high dose of intravenous immunoglobulin (IVIg) in addition to conventional heart failure therapy in patients with idiopathic cardiomyopathy and PVB19 persistence in the heart achieves improvement of cardiac function in conjunction with virus elimination.

Study design: All patients will undergo routine diagnostic work-up (including physical examination, coronary angiogram, transthoracic echocardiogram, blood studies and endomyocardial biopsies (EMB)), treatment and follow-up for their heart failure. Patients will be randomized to either receive IVIg or placebo on top of their standard heart failure regimen.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic cardiomyopathy (LVEF <45%) >6months
* Optimal conventional heart failure medication >3 months.
* PVB19 viral load >200 copies/mcg DNA in endomyocardial biopsies (EMBs).
* Signed informed consent
* Aged between 18 and 75 years

Exclusion Criteria:

* Other causes for heart failure
* Significant coronary artery disease (lesions >70 % stenosis)
* Significant valvular disease
* Untreated hypertension (blood pressure >140mmHg)
* Substance abuse
* Chemotherapy induced
* Significant titer of other cardiotrophic viruses (EV, ADV, HHV6, EBV)
* Pregnancy or lactation
* Systemic diseases such as sarcoidosis, giant cell myocarditis, hemochromatosis, or systemic autoimmune diseases.
* Treatment with any other investigational drug within 7 days before study entry or previous enrolment in this study
* Known with allergic reactions against human plasma or plasma products
* Having an ongoing progressive terminal disease, including HIV infection
* Having renal insufficiency (plasma creatinin >115µmol/L or creatinin clearance <20 ml/min)
* Having an ongoing active disease causing general symptoms e.g. chronic active hepatitis, persistent enterovirus infection with ongoing systemic complaints
* Having detectable anti-IgA antibodies
* Active SLE

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The main study parameter is the change in cardiac ejection fraction presence of the heart from baseline to endpoint. | 6 months

SECONDARY OUTCOMES:
Secondary objectives include changes in presence of cardiotrophic viruses, inflammation , fibrosis, cardiac functional capacity, patient quality of life, other echocardiographic parameters. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: S Heymans, PhD, MD, Principal Investigator — AZM, Maastricht
Locations (1):
- AZM, Maastricht, Netherlands

REFERENCES:
- [Derived] Hazebroek MR, Henkens MTHM, Raafs AG, Verdonschot JAJ, Merken JJ, Dennert RM, Eurlings C, Abdul Hamid MA, Wolffs PFG, Winkens B, Brunner-La Rocca HP, Knackstedt C, van Paassen P, van Empel VPM, Heymans SRB. Intravenous immunoglobulin therapy in adult patients with idiopathic chronic cardiomyopathy and cardiac parvovirus B19 persistence: a prospective, double-blind, randomized, placebo-controlled clinical trial. Eur J Heart Fail. 2021 Feb;23(2):302-309. doi: 10.1002/ejhf.2082. Epub 2021 Jan 7. PMID 33347677